CLINICAL TRIAL: NCT05850039
Title: Study of the Expression of Autophagy Markers in the Myocardium in Patients With Persistent or Permanent Atrial Fibrillation
Acronym: MIPAR-02
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ospedale San Raffaele (Other)
Responsible Party: Principal Investigator, Michele De Bonis, Head of Cardiac Surgery of Advanced and Research Therapies, Ospedale San Raffaele
Other Study IDs: MIPAR-02
Record Dates: First submitted 2023-03-13; First posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-04

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — fragments of posterior left atrial wall measuring between approximately 0.5 x 0.5 cm and approximately 1 x 1 cm and full thickness along the atriotomy incision line near the right pulmonary veins. The sample will be divided into 3 parts: one fixed in 10% buffered formalin for the morphological study by optical microscopy, one frozen in liquid nitrogen for molecular investigations and the last, with dimensions no larger than 1.5 x 1.5 mm and full thickness, fixed in Karnowsky liquid, for electron microscopy study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Study group: Patients with permanent or persistent AFib, undergoing surgical ablation, isolated or concomitant to valve surgery
  Interventions: Other: Sampling
- Mitral surgery control group: Patients undergoing isolated or concomitant mitral valve surgery
  Interventions: Other: Sampling
- Autoptic control group: Autopsy samples in subjects without arrhythmia
  Interventions: Other: Sampling

INTERVENTIONS:
Other: Sampling — Sample collection: a small fragment of atrial wall will be collected

SUMMARY:
Atrial Fibrillation (AFib) is the most common cardiac arrhythmia, causing the loss of the normal and coordinated atrial contractility.

Several studies have demonstrated the existence of some atrial anatomical sites involved in the initiation and maintenance of this arrhythmia, first of all the posterior wall in the area around the outlet of the pulmonary veins. In fact, the existence of a complex of structural and functional modifications has been documented, collectively defined as "structural remodeling" which involve both the cardiomyocyte and the interstitium (the space between the cardiomyocytes) from a histopathological point of view; at the cardiomyocyte level, a loss of sarcomeres in the perinuclear site (myocytolysis), a reduction in the expression of "adult" cellular proteins (e.g. cardiotin and titin) with concomitant re-expression of "fetal" proteins (e.g. muscle actin smooth), as well as a modification of the mitochondrial structure. At the interstitial level, remodeling is characterized by the deposition of fibrous tissue in the interstitium between the muscle bundles and by a reduction in capillary density. Regarding the deposition of collagen fibers, some studies on an experimental model of AFib have shown that the latter is not reversible.

Autophagy is an intracellular process regulated by numerous biochemical signals; it is present at basal levels in most tissues and allows the physiological turnover of the various structural components of the cell, directing them to lysosomal degradation. It can also be stimulated by external signals in unfavorable environmental conditions, such as in the case of pathologies that determine a condition of tissue oxidative stress protracted over time. Experimentally, an excessive activation of the latter has been associated with the early stages of pathological cardiac remodeling in various animal models of cardiovascular diseases and some recent studies have hypothesized that altered levels of autophagy may contribute to the possible mechanisms involved in the generation and maintenance of the remodeling cardiomyocyte and interstitial structure in AFib. The levels of autophagic activity can be evaluated by studying specific markers - such as the Beclin-1 and LC3B proteins - constituents of the autophagic signaling cascade. In the case of LC3B, the "LC3BII/LC3BI" ratio (the processed form of autophagosomal vesicles and the unprocessed form constitutively present at the cytoplasmic level) was used as an autophagy biomarker. Furthermore, some microRNAs (miRNAs) capable of controlling the expression of proteins of the autophagic cascade have been described in the literature. This is the case of miRNA 30a and miRNA 204, respectively, which respectively inhibit the expression of Beclin-1 and of LC3B.

This study aims to investigate from a histo-morphological and molecular point of view the presence of alterations of autophagy mechanisms in patients with persistent or permanent AFib and which correlate these modifications with the degree of structural remodeling present at the level of the left atrial myocardium.

ELIGIBILITY:
Group 1 - Study Inclusion criteria

* Age between 18 and 85 years old
* Permanent or persistent AFib for which the patient undergoes ablation surgery surgery of atrial fibrillation with isolated radiofrequency or associated with possible correction of heart valve disease with or without coronary artery disease Exclusion criteria
* Age < 18 years
* Need for emergency cardiac surgery
* Presence of concomitant systemic inflammatory diseases

Group 2 - Control Inclusion criteria

* Age between 18 and 85 years old
* Sinus rhythm at the time of admission for surgery
* No AFib in history
* Hospitalized for correction of isolated mitral valve disease or associated with correction of other valve diseases Exclusion criteria
* Age < 18 years
* Need for surgical coronary revascularization
* Need for emergency cardiac surgery
* Presence of concomitant systemic inflammatory diseases

Group 3 - Autoptic control Inclusion criteria

* Age between 18 and 85 years old Exclusion criteria
* No signs of post-mortal tissue decomposition assessed by histological examination
* Documented history of arrhythmias, valvular dysfunction, atherosclerosis of the coronary arteries, previous myocardial infarctions, foci of myocardial fibrosis greater than 2 mm on histology, presence of inflammatory cells in the interstitium, sarcoidosis, amyloidosis, chronic inflammatory lung diseases and connective tissue diseases.

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Group 1 - Study
Sampling Method: Non-Probability Sample
Enrollment: 81 (Estimated)
Dates: Start 2019-04-09 (Actual); Primary Completion 2024-04-09 (Estimated); Study Completion 2024-06-09 (Estimated)

PRIMARY OUTCOMES:
Beclin-1 and LC3B levels in blood | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No